CLINICAL TRIAL: NCT01926431
Title: The Effects of High Intensity Exercise on Neural Responses to Images of Food
Brief Title: Effects of Intense Exercise on Neural Responses to Food.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Principal Investigator, Daniel Crabtree, Principal Investigator, University of Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: fMRI Study; ERN_09-586 (Registry Identifier: University of Birmingham)
Record Dates: First submitted 2013-08-20; First posted 2013-08-21 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Neural Responses; Appetite Hormones; Subjective Appetite Sensations
MeSH Terms: interventions — Exercise; RE1-silencing transcription factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): 60 minutes of high intensity treadmill running
  Interventions: Other: Exercise
- Rest (Experimental): 60 minutes of seated rest (control trial)
  Interventions: Other: Rest

INTERVENTIONS:
Other: Exercise
  Arms: Exercise
Other: Rest
  Arms: Rest

SUMMARY:
The primary aim of this study was to determine the effects of an acute bout of high intensity exercise on the brains response to viewing pictures of food using functional magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
It is clear that intense exercise impacts on peripheral appetite regulation, however very little is known about the impact of high-intensity exercise on central appetite regulation. This study aimed to investigate the effects of high-intensity exercise on both central and peripheral responses to images of food. Functional magnetic resonance techniques were used to assess the brains response to images of high and low calorie foods, following a short bout of high-intensity exercise. Appetite hormone concentrations were also measured. It was hypothesized that, due to the known effects of high-intensity exercise on appetite regulatory hormones and subjective appetite ratings, the activation of reward-related brain regions to visual food cues would be modulated following intense physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smokers, free from cardiovascular disease and metabolic disease, no medication, participated in moderate/vigorous physical activity (>2 hours per week)

Exclusion Criteria:

* Smokers, history of cardiovascular/metabolic disease, low physical activity levels, inability to participate in fMRI scanning sessions including contraindications to MRI

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Neural responses following exercise and rest | Ten minutes post-exercise/rest
  Volunteers completed an fMRI assessment following 60 minutes of intense exercise and 60 minutes of rest on two separate occasions.

SECONDARY OUTCOMES:
Appetite hormones | Blood samples taken at baseline, following exercise/rest, prior to the fMRI assessment and immediately following the fMRI assessment
  Blood samples were taken using a cannula system for both trials. Concentrations of appetite regulating hormones were measured from plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Blannin, PhD, Principal Investigator — University of Birmingham
Locations (1):
- Birmingham University Imaging Centre, Birmingham, Midlands, United Kingdom

REFERENCES:
- [Derived] Crabtree DR, Chambers ES, Hardwick RM, Blannin AK. The effects of high-intensity exercise on neural responses to images of food. Am J Clin Nutr. 2014 Feb;99(2):258-67. doi: 10.3945/ajcn.113.071381. Epub 2013 Dec 4. PMID 24305681